CLINICAL TRIAL: NCT07083557
Title: Routine Validation and Reproducibility Testing of Laboratory Assays and Research Techniques Used for Endocrine, Cardiometabolic, and Musculoskeletal Disorder Research (VALD)
Acronym: VALD
Status: Recruiting | Type: Observational
Sponsor: Bettina Mittendorfer (Other)
Responsible Party: Sponsor-Investigator, Bettina Mittendorfer, Senior Associate Dean for Research; Professor, Medicine & Nutrition; NextGen Director of Clinical and Translational Sciences Unit, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Other Study IDs: 2127348
Record Dates: First submitted 2025-05-30; First posted 2025-07-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Obesity-related Medical Conditions; Diabetes; Atherosclerotic Disease; Heart Failure; MASH; Sarcopenia; Osteoporosis; Hyperparathyroidism; Hypoparathyroidism; Ischemic Heart Disease; Cystic Fibrosis (CF); Chronic Kidney Disease(CKD); Osteopenia; Cachexia
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Heart Failure; Sarcopenia; Osteoporosis; Hyperparathyroidism; Hypoparathyroidism; Myocardial Ischemia; Cystic Fibrosis; Renal Insufficiency, Chronic; Bone Diseases, Metabolic; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endothelial cell collection — Participants may opt to have testing performed including blood sampling, urine sampling, intravenous catheter placement with endothelial cell collection, oral glucose tolerance test, consuming a test meal, having imaging performed such as MRI, DEXA, MRS, having adipose (fat) or muscle biopsies, or non-invasive endothelial function testing to investigate use of different assays, different sample treatment approaches to determine optimal conditions that produce the most accurate and reproducible results, and/or repeat testing on different days or with different equipment that measures the same variable.

SUMMARY:
The purpose of this research study is to validate (check the accuracy of) laboratory assays, intravenous catheter insertion, and equipment or devices and their reproducibility, which is necessary to perform high quality research on chronic diseases, nutrition, and metabolism (the process by which a substance is handled in the body) at the University of Missouri. As technology changes and uses new testing methods, it is necessary to compare results from old tests, equipment and devices and new tests, equipment, or devices and the reproducibility of these measurements to make sure the results are accurate. Reproducibility means performing the same test more than once to see if the same results can be achieved each time. This study will look at the validation and reproducibility of tests and laboratory assays in participants who are healthy or affected by relevant endocrine, cardiometabolic, and musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤100 years of age
* body mass index ≥16.0 and ≤60 kg/m2

Exclusion Criteria:

* <18 and >100 years of age
* body mass index <16.0 or >60 kg/m2
* allergies, intolerances, or dietary restrictions to meal ingredients, vegans or vegetarians
* use of medications or dietary supplements (e.g., anti-inflammatories, immune modulators, etc) that could interfere with the particular assay/techniques being evaluated
* engaged in regular structured exercise >150 min per week unless needed for validation of the assay/technique being evaluated
* significant organ system dysfunction or diseases, except those that are sought for validation of the assay/technique being evaluated
* alcohol use disorder as defined by the National Institute of Alcohol Abuse and Alcoholism or use of controlled substances unless alcohol use disorder is required for validation of the assay/technique being evaluated
* pregnant women, persons who smoke, prisoners, and inability to grant voluntary informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: convenience population of volunteers in mid-Missouri region
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the validity and reproducibility of insulin results in the laboratory environment | through study completion, up to 6 months
  Comparison of insulin results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Validation and reproducibility testing for endothelial cell collection | through study completion, up to 6 months
  endothelial cell quantity collected
Validation and reproducibility testing for mixed meal ingestion | through study completion, up to 6 months
  palatability of meal type (protein concentration, carbohydrate concentration) as measured by amount of meal consumed
Evaluation of the validity and reproducibility of urinalysis results in the laboratory environment | through study completion, up to 6 months
  Comparison of urinalysis results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Validation and reproducibility testing for glucose tolerance testing | through study completion, up to 6 months
  glucose levels (mg/dL) at various time points including fasting, random, and postprandial
Validation and reproducibility testing for DEXA | through study completion, up to 6 months
  body composition analysis (percentage fat and muscle)
Validation and reproducibility testing for MRI | through study completion, up to 6 months
  body composition analysis (percentage fat and muscle)
Validation and reproducibility testing for MRS | through study completion, up to 6 months
  body composition analysis (percentage fat and muscle)
Validation and reproducibility of vascular (endothelial) function test | through study completion, up to 6 months
  non-invasive vascular function test (measured using EndoPat machine)
Validation and reproducibility of adipose (fat) tissue biopsy | through study completion, up to 6 months
  microscopic characteristics of tissue collected
Validation and reproducibility testing of muscle tissue biopsies | through study completion, up to 6 months
  microscopic characteristics of tissue collected
Evaluation of the validity and reproducibility of C-peptide results in the laboratory environment | through study completion, up to 6 months
  Comparison of C-peptide results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of glucagon results in the laboratory environment | through study completion, up to 6 months
  Comparison of glucagon results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of free fatty acid level results in the laboratory environment | through study completion, up to 6 months
  Comparison of free fatty acid level results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of glucose results in the laboratory environment | through study completion, up to 6 months
  Comparison of glucose results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of ketone body results in the laboratory environment | through study completion, up to 6 months
  Comparison of ketone body results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of cytokine results in the laboratory environment | through study completion, up to 6 months
  Comparison of cytokine results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of adipokine results in the laboratory environment | through study completion, up to 6 months
  Comparison of adipokine results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of lipid profile results in the laboratory environment | through study completion, up to 6 months
  Comparison of lipid profile results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine calcium results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine calcium results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine magnesium results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine magnesium results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine phosphorous results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine phosphorous results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine sodium results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine sodium results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine oxalate results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine oxalate results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations
Evaluation of the validity and reproducibility of urine citrate results in the laboratory environment | through study completion, up to 6 months
  Comparison of urine citrate results across assays (methods of measuring) to evaluate the validity and reproducibility in the basic science laboratory environment across healthy and disordered populations

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No